CLINICAL TRIAL: NCT03155815
Title: Dementia Population Risk Tool (DemPoRT): A Predictive Algorithm for Assessing Dementia Risk in the Community Setting
Brief Title: Assessing Dementia Risk in the Community: The Dementia Population Risk Tool
Acronym: DemPoRT
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Institute for Clinical Evaluative Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: CIHR FRN 142237
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Derivation Cohort: Eligible respondents to the combined 2001, 2003, 2005 and 2007 Canadian Community Health Surveys, conducted by Statistics Canada.
- Validation Cohort: Eligible respondents to the 2008/2009 Canadian Community Health Survey.

SUMMARY:
The purpose of this study is to develop and validate the Dementia Population Risk Tool (DemPoRT) algorithm to predict dementia incidence in the population setting.

DETAILED DESCRIPTION:
The burden of disease from dementia is a growing global concern as incidence increases exponentially with age and average life expectancy has been increasing around the world. Planning for an aging population requires reliable projections of future dementia prevalence and resource requirements, however, existing population projections are simple and have poor predictive accuracy. The Dementia Population Risk Tool (DemPoRT) will predict incidence of dementia in the population setting using multivariable modeling techniques.

The derivation cohort will consist of elderly Ontario respondents of Canadian Community Health Survey (CCHS) (2001, 2003, 2005, 2007; approximately 19 000 males and 25 000 females). Pre-specified predictors include sociodemographic, general health, behavioral, functional and health condition variables. Incident dementia will be identified through individual linkage of survey respondents to population-level administrative health care databases. Using time of first dementia capture as the primary outcome and death as a competing risk, sex-specific proportional hazards regression models will be estimated. The 2008/2009 CCHS survey be used for validation (approximately 4 600 males and 6 300 females). Overall calibration and discrimination will be assessed as well as calibration within predefined subgroups of importance to clinicians and policy makers.

ELIGIBILITY:
Inclusion Criteria:

* Respondents to the Canadian Community Health Surveys

Exclusion Criteria:

* Less than 55 years of age at survey administration
* Prior history of dementia
* Not eligible for Ontario's universal health insurance program

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The derivation cohort will be eligible respondents to the combined 2001, 2003, 2005 and 2007 Canadian Community Health Surveys, conducted by Statistics Canada. The validation cohort will consist of respondents to the 2008/2009 survey.
Sampling Method: Probability Sample
Enrollment: 75460 (Actual)
Dates: Start 2000-09 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Dementia capture in administrative data | Up to 13 years
  Identification of incident dementia in administrative data using a validated case ascertainment definition, supplemented by dementia codes captured on home care and long-term care assessments

CONTACTS AND LOCATIONS:
Overall Officials: Peter Tanuseputro, Principal Investigator — Ottawa Hospital Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher S, Hsu A, Mojaverian N, Taljaard M, Huyer G, Manuel DG, Tanuseputro P. Dementia Population Risk Tool (DemPoRT): study protocol for a predictive algorithm assessing dementia risk in the community. BMJ Open. 2017 Oct 24;7(10):e018018. doi: 10.1136/bmjopen-2017-018018. PMID 29070641